CLINICAL TRIAL: NCT04916119
Title: A Phase I, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of IBI323 in Participants With Advanced Malignancies
Brief Title: Study of IBI323 in Patients With Advanced Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI323A101
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI323 (Experimental): Phase Ia enrolls patients with advanced malignancies. Phase Ib cohort A enrolls patients with NSCLC(IO-refractory), cohort B NSCLC(IO-naive), cohort C NSCLC(PD-L1 TPS≥1%), cohort D ES-SCLC or neuroendocrine tumors, cohort E MPM, cohort F UC, cohort G nccRCC, cohort H HCC, cohort I NPC, cohort J CC or HNSCC, cohort K GC or GEJC with HER2 negative, cohort L TNBC
  Interventions: Drug: IBI323

INTERVENTIONS:
Drug: IBI323 — In phase Ia study, seven dose levels of IBI323 (0.03, 0.1, 0.3, 1, 3, 10 and 20mg/kg) will be evaluated. The DLT observation period is 28 days. IBI323 is administered by iv infusion day 1 of every 14 days. After dose escalation stage completed, two dose levels (10mg/kg and 20mg/kg) will be expanded to 20 patients each. In Phase Ib study, IBI323 is administered RP2D by iv infusion day 1 of every 14 days. IBI323 and chemotherapy will be administrated in cohort C and cohort K

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and efficacy of IBI323(anti-LAG-3/PD-L1) or in combination with chemotherapy in participants with advanced malignancies. Another purpose is to determine the pharmacokinetics,pharmacodynamics and immunogenicity of IBI323

ELIGIBILITY:
Inclusion Criteria:

1. Phase Ia Patients with locally advanced, recurrent or metastatic solid tumors who have failed standard treatment Phase Ib cohort A Patients with IO-refractory advanced NSCLC cohort B Patients with IO-naive advanced NSCLC who have failed standard treatment cohort C Patients with advanced NSCLC who have no prior treatment and PD-L1 TPS≥1% cohort D Patients with ES-SCLC or G3 neuroendocrine tumors who have failed standard treatment cohort E Patients with advanced MPM who have failed standard treatment cohort F Patients with advanced UC who have failed standard treatment cohort G Patients with advanced nccRCC who have failed standard treatment cohort H Patients with advanced HCC who have failed standard treatment cohort I Patients with advanced NPC who have failed standard treatment cohort J Patients with advanced CC or HNSCC who have failed standard treatment cohort K Patients with advanced GC or GEJC with HER2 negative who have no prior treatment cohort L Patients with advanced TNBC who have failed standard treatment
2. Able to understand and willing to sign the ICF.
3. 18 to 75 years old.
4. Life expectancy at least 12 weeks.
5. At least 1 measurable lesion per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate organ and bone marrow functionAdequate organ and bone marrow function.

Exclusion Criteria:

1. Prior treatment with any anti- LAG-3 antibody.
2. Prior immunotherapy treatment for Stage Ia extension cohort ( immunotherapy untreated) and Stage Ib cohort B-L
3. Any investigational drugs received within 4 weeks prior to the first study treatment.
4. Receive the last dose of anti-tumor therapy within 4 weeks before the first dose of study therapy.
5. Symptomatic CNS metastasis.
6. History of autoimmune disease , present active autoimmune disease or inflammatory diseases
7. Pregnant or nursing females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-12-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 24 months
  To evaluate the safety and tolerability of IBI323 [Adverse events (AEs), treatment-related AE (TRAE), immune-related AEs (irAE), serious adverse event (SAE), dose-limiting toxicity (DLT) assessed by CTCAE v5.0]

SECONDARY OUTCOMES:
Investigator Assessments of Overall Response Rate(ORR) | 24 months
  RECIST v1.1 will be used to determine ORR by investigator
Disease Control Rate(DCR) | 24 months
  RECIST v1.1 will be used to determine DCR by investigator
PFS (progression-free survival) | 24 months
  RECIST v1.1 will be used to determine PFS by investigator
Anti-drug antibody (ADA) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shang Hai Pulmonary Hospital, Shanghai, Shanghai Municipality, China